CLINICAL TRIAL: NCT02851147
Title: Slit Lamp Model SL-D-301 and DC-4 Digital Camera Attachment
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: TOPCON-007-2016
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Ocular Images

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Any Willing and Able Person for Ocular Imaging: Any Willing and Able Person for Ocular Imaging
  Interventions: Device: SL-D301; Device: DC-4; Device: SL-3G

INTERVENTIONS:
Device: SL-D301 — Slit Lamp
Device: DC-4 — Digital Camera Attachment
Device: SL-3G — Slit Lamp

SUMMARY:
The purpose of the evaluation is to confirm operability and usability of the SL-D301 Slit Lamp and the DC-4 digital camera attachment by conducting a usability evaluation and subsequently submitting a questionnaire and hold an interview with the operator.

Of special interest for the study is to confirm whether the illumination level of SL-D301 is enough to perform an eye exam since the maximum illumination level on the SL-D301 is lower than other existing Topcon digital ready slit lamps due to regulations that limit the maximum light intensity on the human eye. The SL-D301 will be compared against the predicate device SL-3G.

DETAILED DESCRIPTION:
An eye care professional familiar with the use of slit lamps and experienced with other Topcon and other manufacturer's slit lamps will evaluate operability and usability of SL-D301 and DC-4 digital camera attachment instrument performing routine eye examinations and image capture on volunteer subjects using above mentioned instruments. Similar evaluations will be performed with the SL-3G Slit Lamp and a comparative evaluation will be drawn between the two instruments. At the end of the evaluation, the evaluator will be presented with a questionnaire on specific points regarding the performance and features of the instruments and interviewed. The responses will then be evaluated by Topcon.

ELIGIBILITY:
Inclusion Criteria:

* Any Willing Subject

Exclusion Criteria:

* Subjects unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of a maximum number of 30 volunteer subjects consenting to undergo a slit lamp eye exam and to have digital images of their eyes obtained with the DC-4 and the SL-D301.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Image Comparison of DC-4 to the SL-D301 | 1 Hour

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Almiron, Study Chair — Topcon Corporation
Locations (1):
- Glassman Eye Associates, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided